CLINICAL TRIAL: NCT04216043
Title: Milk Matters in Malnutrition, is it the Lactose or Dairy Protein?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Project Peanut Butter, Sierra Leone (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201912091
Record Dates: First submitted 2019-12-23; First posted 2020-01-02 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Malnutrition, Child
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The RUSF food products are very similar in appearance and texture; thus, subjects and caretakers will be blinded. The investigators making the clinical assessments will not have information as to specialized food product assignment of the subject, and will remain blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RUSF skimmed milk powder (Experimental): RUSF will provide 75 kcal/kg/day (314 kJ/kg/day) and full daily doses of vitamins and micronutrients. Caregivers will instruct caregivers to feed the supplement only to the enrolled child, to feed it in addition to their usual diet, and to use daily portions.
  Interventions: Dietary Supplement: RUSF skimmed milk powder
- RUSF milk protein concentrate and sucrose (Experimental): RUSF will provide 75 kcal/kg/day (314 kJ/kg/day) and full daily doses of vitamins and micronutrients. Caregivers will instruct caregivers to feed the supplement only to the enrolled child, to feed it in addition to their usual diet, and to use daily portions.
  Interventions: Dietary Supplement: RUSF milk protein concentrate and sucrose
- RUSF soy protein and whey permeate (Experimental): RUSF will provide 75 kcal/kg/day (314 kJ/kg/day) and full daily doses of vitamins and micronutrients. Caregivers will instruct caregivers to feed the supplement only to the enrolled child, to feed it in addition to their usual diet, and to use daily portions.
  Interventions: Dietary Supplement: RUSF soy protein and whey permeate
- RUSF soy and sucrose (Experimental): RUSF will provide 75 kcal/kg/day (314 kJ/kg/day) and full daily doses of vitamins and micronutrients. Caregivers will instruct caregivers to feed the supplement only to the enrolled child, to feed it in addition to their usual diet, and to use daily portions.
  Interventions: Dietary Supplement: RUSF soy and sucrose

INTERVENTIONS:
Dietary Supplement: RUSF skimmed milk powder — ready-to-use supplementary foods 75 kcal/kg/day (314 kJ/kg/day) and full daily doses of vitamins and micronutrients
  Arms: RUSF skimmed milk powder
Dietary Supplement: RUSF milk protein concentrate and sucrose — ready-to-use supplementary foods 75 kcal/kg/day (314 kJ/kg/day) and full daily doses of vitamins and micronutrients
  Arms: RUSF milk protein concentrate and sucrose
Dietary Supplement: RUSF soy protein and whey permeate — ready-to-use supplementary foods 75 kcal/kg/day (314 kJ/kg/day) and full daily doses of vitamins and micronutrients
  Arms: RUSF soy protein and whey permeate
Dietary Supplement: RUSF soy and sucrose — ready-to-use supplementary foods 75 kcal/kg/day (314 kJ/kg/day) and full daily doses of vitamins and micronutrients
  Arms: RUSF soy and sucrose

SUMMARY:
This study is to look at the types of sugar and protein composition in the treatment of moderate acute malnutrition and its effects on gut health. The study will use 4 different types of ready to use supplementary foods to see which one if any has better recovery rate along with looking into the gut health. Children will be treated using one food for up to 12 weeks. A subset of about 400 will be tested for intestinal permeability using the dual sugar test.

ELIGIBILITY:
Inclusion Criteria:

* MUAC < 12.5 cm and ≥ 11.5 cm without bipedal oedema

Exclusion Criteria:

* If they are involved in another research trial
* in another supplemental feeding program
* debilitating illness
* history of peanut or milk allergy

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1102 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
% lactulose excretion after 4 weeks of supplementary feeding | 4 weeks
  This will only be assessed in children with higher-risk (MUAC < 12 cm) MAM at baseline.
  %L measured in the urine relative to the amount ingested will be calculated. %L will be categorized as normal (<0.2%) and abnormal (>0.2)
16S rRNA relative abundance of bacterial taxa after 4 weeks of supplementary feeding | 4 weeks
  This will only be assessed in children with higher-risk (MUAC < 12 cm) MAM at baseline

SECONDARY OUTCOMES:
Rate of weight gain (g/kg/d) | up to 12 weeks of treatment
  Changes in weight relative to baseline weight
Rate of length gain (mm/week) | up to 12 weeks of treatment
  Changes in linear growth
Final mid-upper arm circumference | up to 12 weeks of treatment
  Use the mid-upper are circumference at the visit when outcome was reached
Proportion with %L < 0.20 | 4 weeks
  Percentage of children with %L excreted < 0.20
16S rRNA beta-diversity at week 4 | 4 weeks
  Looking at the 16S configuration in stool samples collected
16S rRNA alpha-diversity at week 4 | 4 weeks
  Several metrics of alpha diversity will be assessed, including Shannon's index
Rate of recovery from moderate acute malnutrition | up to 12 weeks of treatment
  Recovery is when a participant reaches a Mid-Upper Arm Circumference of 12.5cm or better
Rate of deteriorating to severe acute malnutrition or death | up to 12 weeks of treatment
  Severe acute malnutrition defined by MUAC < 11.5 cm or development of nutritional edema
Sub-group analysis of %L and 16S rRNA outcomes among children not receiving breastfeeding at baseline vs. those being breastfeed at baseline | 4 weeks
  Anthropometric, %L and 16s rRNA outcomes (relative abundance, alpha-diversity, beta-diversity) will be compared between study foods among those who are reported to be breastfeeding vs. those who are not
Sub-group analysis of anthropometric outcomes among children with MUAC < 12 cm vs. >= 12 cm at baseline | up to 12 weeks of treatment
  Rate of weight change, length change, final MUAC, recovery, SAM, and death will be compared between the study foods among children with baseline MUAC < vs. >=12 cm.
Metabolomic feature abundance in the 4 dietary groups | After 4 weeks of supplementary feeding
  Metabolomic feature abundance in the 4 dietary groups, as determined by untargeted metabolomics in 200 randomly selected children with MUAC < 12.1 cm on enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Mark Manary, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Project Peanut Butter Factory, Freetown, Sierra Leone

REFERENCES:
- [Background] Black RE, Allen LH, Bhutta ZA, Caulfield LE, de Onis M, Ezzati M, Mathers C, Rivera J; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: global and regional exposures and health consequences. Lancet. 2008 Jan 19;371(9608):243-60. doi: 10.1016/S0140-6736(07)61690-0. No abstract available. PMID 18207566
- [Background] Caulfield LE, de Onis M, Blossner M, Black RE. Undernutrition as an underlying cause of child deaths associated with diarrhea, pneumonia, malaria, and measles. Am J Clin Nutr. 2004 Jul;80(1):193-8. doi: 10.1093/ajcn/80.1.193. PMID 15213048
- [Background] Shankar AH. Nutritional modulation of malaria morbidity and mortality. J Infect Dis. 2000 Sep;182 Suppl 1:S37-53. doi: 10.1086/315906. PMID 10944483
- [Background] Matilsky DK, Maleta K, Castleman T, Manary MJ. Supplementary feeding with fortified spreads results in higher recovery rates than with a corn/soy blend in moderately wasted children. J Nutr. 2009 Apr;139(4):773-8. doi: 10.3945/jn.108.104018. Epub 2009 Feb 18. PMID 19225128
- [Background] Nackers F, Broillet F, Oumarou D, Djibo A, Gaboulaud V, Guerin PJ, Rusch B, Grais RF, Captier V. Effectiveness of ready-to-use therapeutic food compared to a corn/soy-blend-based pre-mix for the treatment of childhood moderate acute malnutrition in Niger. J Trop Pediatr. 2010 Dec;56(6):407-13. doi: 10.1093/tropej/fmq019. Epub 2010 Mar 23. PMID 20332221
- [Derived] Son M, Laury ML, Stephenson KB, May T, Hendrixson DT, Koroma AS, Ngegbai AS, Song JH, Naskidashvili N, Goo YA, Manary MJ. The Impact of Milk on Gut Permeability, Fecal 16S rRNA Gene Microbiota Profiling, and Fecal Metabolomics in Children with Moderate Malnutrition in Sierra Leone: A Double-Blind, Randomized Controlled Trial. Am J Clin Nutr. 2024 Nov;120(5):1114-1124. doi: 10.1016/j.ajcnut.2024.09.018. Epub 2024 Sep 21. PMID 39307188